CLINICAL TRIAL: NCT06339229
Title: Association Between Postoperative New-onset Proteinuria and Adverse Outcomes: a Retrospective Cohort Study.
Brief Title: Postoperative New-onset Proteinuria and Adverse Outcomes.
Status: Completed | Type: Observational
Sponsor: Yaozhong Kong (Other)
Responsible Party: Sponsor-Investigator, Yaozhong Kong, Professor, First People's Hospital of Foshan
Organization: First People's Hospital of Foshan (Other)
Other Study IDs: FSYYY-2024-12
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Surgery; Proteinuria; Mortality
MeSH Terms: conditions — Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- surgery patients
  Interventions: Other: proteinuria

INTERVENTIONS:
Other: proteinuria — dipstick proteinuria values negative, trace, 1+, and ≥2+

SUMMARY:
We aimed to assess the association between postoperative new-onset proteinuria, all-cause mortality, and decline in kidney function in Chinese people who underwent surgery. The exposure variable was the dipstick proteinuria values from the initial postoperative urinalysis within 30 days after surgery, categorized as negative, trace, 1+, and ≥2+. The primary outcome was 30-day mortality. The secondary outcomes included 1-year mortality and composite kidney outcome assessed using the postoperative estimated glomerular filtration rate.

ELIGIBILITY:
Inclusion Criteria:

* surgery patients

Exclusion Criteria:

* kidney or urinary surgery
* missing urinalysis results
* dipstick proteinuria indicated a value of "≥ trace" at least once preoperatively
* with dialysis, end-stage renal disease, or with urinary tract infection at baseline
* missing follow-up information

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Using the International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM) codes, participants aged ≥16 years who underwent surgery from January 2000 to December 2022 were included.
Sampling Method: Non-Probability Sample
Enrollment: 2983899 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
mortality | 30-day